CLINICAL TRIAL: NCT00983307
Title: A Phase II Study of Erlotinib (Tarceva) and Hypofractionated Thoracic Radiotherapy for Patients With Advanced or Inoperable Non-Small-Cell Lung Cancer
Brief Title: A Study of Erlotinib Plus Radiotherapy (RT) for Patients With Advanced or Inoperable Non-Small-Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09G.104; 2008-43 (Other: CCRRC); OSI4327s (Other: Genentech); JT 1381 (Other: JeffTrial Number)
Record Dates: First submitted 2009-09-22; First posted 2009-09-24 (Estimated); Results first posted 2018-01-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Carcinoma, Non-small-cell Lung
Keywords: Radiation; Erlotinib; Tarceva
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Radiation Dose Hypofractionation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Erlotinib and radiotherapy (Experimental): Patients will be treated with Erlotinib and hypofractionated radiotherapy.
  Interventions: Drug: Erlotinib; Radiation: Hypofractionated Radiotherapy

INTERVENTIONS:
Drug: Erlotinib — Patients will receive Tarceva, 150 mg daily on days -5 through -1 days and will start a course of hypofractionated thoracic RT on Day 1. RT will be administered daily on weekdays (Monday-Friday) and not on weekends or holidays. Tarceva administration will be continued daily during RT (also on weekends/holidays when RT is not given) and after RT will be continued daily as maintenance therapy until death or disease progression.
  Other Names: Erlotinib (OSI-774); Tarceva
Radiation: Hypofractionated Radiotherapy — Patients undergo hypofractionated thoracic RT 5 days a week for approximately 2.5 weeks beginning on day 0. Patients also receive erlotinib hydrochloride PO daily beginning on day -5 and continuing for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Other Names: Radiation Therapy; RT

SUMMARY:
It is generally accepted that the presence of chronically hypoxic cells, or tumor cells which do not receive enough oxygen as a result of tumor growth, may be an important cause of resistance to radiation therapy (RT) and resultant tumor recurrence, particularly in large tumors such as advanced non-small-cell lung cancer (NSCLC). Therefore, delivering a higher RT dose, as is done with hypofractionated RT, to the tumor may result in higher success rate.

Erlotinib (Tarceva, previously known as OSI-774) is an orally active, potent, selective inhibitor of the Epidermal Growth Factor Receptor (EGFR) tyrosine kinase. A recently completed trial has shown that Erlotinib as a single agent significantly improves the survival of patients with incurable Stage IIIb/IV NSCLC who have failed standard therapy for advanced or metastatic disease. Therefore, Erlotinib is an approved medication for second-line therapy in lung cancer following prior chemotherapy.

This is a Phase II clinical research study to assess the efficacy and toxicity of hypofractionated radiation therapy in combination with Erlotinib in patients with locally advanced or inoperable non-small-cell lung cancer (NSCLC).

The investigators' hypothesis is that the addition of erlotinib to RT will result in radiosensitization, therefore increasing the likelihood of local tumor control over RT alone. Maintenance erlotinib upon RT completion will result in further tumor growth inhibition, both systemically and locally, lengthening disease-free survival and overall survival.

DETAILED DESCRIPTION:
Hypothesis/Rationale: Lung cancer is the number one cause of cancer-related mortality in both men and women in the United States, with over 170,000 cases diagnosed annually. The overall 5-year survival rate remains 14% despite decades of clinical research. Thoracic RT is the standard treatment for locally advanced (Stage III) NSCLC, in combination with chemotherapy in favorable patients. Metastatic lung cancer (Stage IV) is treated with systemic chemotherapy, with the addition of RT for palliation of tumor symptoms. Most lung cancers present as large tumors, measuring 2 to 7 cm in largest dimension. It is therefore not difficult to understand that only 16% of patients experience a complete resolution of their irradiated tumors within 3 months following a course of standard fractionated (2.0 Gy daily) RT and chemotherapy.

From basic principles advocated by Fletcher, it is thought that standard fractionated RT doses up to 100.0 Gy may be necessary to sterilize tumors of the size frequently encountered in clinical practice. Tumor control probability for bronchogenic carcinoma can be estimated to be 10% for tumors of greater than 4 cm at a dose of 80.0 Gy, with an assumption, that an average-size lung cancer may require doses beyond 100.0 Gy standard fractionated to have a 50% to 80% probability of controlling the tumor. This has been demonstrated in the "stereotactic radioablation" approach to patients with the medically inoperable Stage I NSCLC, in whom 20 Gy per fraction to a total of 60 Gy (a BED equivalent of >100 Gy) resulted in an excellent local control of >90% (Timmerman R et al, 2006; Onishi H et al, 2007).

Hypofractionated RT: It is generally accepted that the presence of chronically hypoxic cells within tumors may be an important cause of radioresistance and resultant local failure in radiotherapy, particularly in large solid tumors such as locoregionally advanced NSCLC. In-vitro experiments indicated that the dose needed to kill severely hypoxic cells is on the order of 2 or 3 times the dose needed for oxic cells. Therefore, delivering a higher RT dose to the tumor may result in higher tumor cell kill and improved local control. One of the approaches to increase RT dose is to use hypofractionated RT, which not only increases the dose, but also reduces the overall treatment time. The radiobiological rationale for hypofractionated RT was described by Mehta et al (Mehta et al, 2001). Based on these theoretical assumptions, University of Wisconsin has recently completed a dose escalation study of progressively increasing fraction sizes in thoracic RT for lung cancer. Such larger RT fraction sizes may require "tighter" radiation fields (to achieve reliable normal-tissue sparing) and improved precision of RT delivery, something that is afforded by the SBF (Stereotactic Body Frame) immobilization and daily CT scan based image verification of tumor position. More experiences have been reported in the literature on hypofractionated regimens for lung cancer. Japanese investigators (Nagata Y et al, 2002) treated 40 patients with T1-T3N0 tumors or lung metastases with 10-12 Gy per fraction to a total of 40-48 Gy. No pulmonary (or other) complications >Grade 2 were observed and the local control was 100% in the subgroup of primary lung tumors. Another group from Japan (Onimaru R et al, 2003) reported on 45 patients with primary lung tumors up to 6cm receiving 7.5 Gy per fraction to 60 Gy (lesions <3cm) or 6 Gy per fractions to 48 Gy (lesions 3-6cm). One patient with a central tumor died of a radiation-induced ulcer in the esophagus. One patient with a peripheral lesion experienced Grade 2 chest wall pain. The 3-year local control rate was 80%. No adverse respiratory events were noted.

The "ultimate" hypofractionated RT regimen of 60 Gy given in 3 fractions of 20 Gy each has been demonstrated to be feasible and highly effective in patients with medically inoperable Stage I NSCLC tumors measuring up to 7 cm and located outside the central airways (Timmerman et al, 2006). However, the same regimen was associated with a high incidence of severe toxicity if applied to central airway. Since most tumors in patients with Stage III and IV NSCLC are located centrally, a novel hypofractionated regimen needs to be developed specifically for them.

In our institution we have completed a Phase I/II investigator-initiated trial of dose-escalated hypofractionated RT given concurrently with Gefitinib (Iressa) with Gefitinib continued after RT completion until progression or toxicity. Three RT dose levels are applied: 4.2 Gy in 10 fractions to 42 Gy; 4.2 Gy in 12 fractions 50.4 Gy and 4.2 Gy in 15 fractions to 63 Gy. Eligible pts are those with either Stage III or IV NSCLC who needed thoracic RT and could not receive chemotherapy. No selection by the EGFR receptor status has been applied. A total of 12 patients have been enrolled. Main toxicities were pulmonary (1 grade 2 pneumonitis; 1 grade 3 infectious pneumonia; 1 grade 4 pneumonitis). There was 1 grade 3 abdominal pain. One patient (with thoracic tumor controlled) died due to the late radiation-esophageal toxicity (tracheo-esophageal fistula in a setting of pre-existing esophageal diverticula) at 12 months from RT. Only one patient experienced local progression of the irradiated tumor, which is very encouraging and may support the hypothesis of the radiosensitizing effect of the EGFR inhibitors. As of now, median survival time for all 12 enrolled patients is 9 months (range: 1-26 mo) from the time of initiating Gefitinib, which is an encouraging result in mostly pretreated patients, many with metastatic disease (Werner-Wasik et al, oral presentation, First ESMO/IASLC European Meeting on Lung Cancer, Geneva, Switzerland, April 2008).

Since Gefitinib is not available now for wider use, we are proposing a study of erlotinib with hypofractionated RT in a Phase II setting with the main objective of assessing efficacy of such a combination. There is no direct evidence that patients receiving concurrent EGFR inhibitors and RT need to be pre-selected with regard to the EGFR status. In a recent study (Bentzen SM et al, 2005), positive immunohistochemical staining for EGFR status was associated with a benefit in locoregional control in patients with head and neck cancer receiving CHART (continuous hyperfractionated accelerated radiotherapy), but the EGFR status had no effect on survival or rate of distant metastases. Therefore, we propose to investigate the EGFR status in all eligible patients, but to treat them without selection for the EGFR status.

Tarceva (previously known as OSI-774) is an orally active, potent, selective inhibitor of the EGFR tyrosine kinase. Early clinical data with Tarceva indicate that the compound is generally safe and well tolerated at doses that provide the targeted effective concentration based on nonclinical experiments. A recently completed, randomized, double-blind, placebo-controlled trial (BR.21) has shown that Tarceva as a single agent significantly improves the survival of patients with incurable Stage IIIb/IV NSCLC who have failed standard therapy for advanced or metastatic disease (Shepherd F et al, 2000 and 2005). In a Phase II clinical trial (Jackman D et al, 2007) of 80 chemotherapy-naive patients >70 years of age with advanced non-small cell lung cancer who received erlotinib as first-line therapy, an encouraging median survival time (MST) of 10.9 months was reported, with the presence of EGFR mutations strongly correlated with disease control and survival.

In summary, a combination of erlotinib with hypofractionated thoracic RT has the potential to significantly improve local tumor control in patients with non-small-cell lung cancer, based on theoretical considerations of EGFR inhibition, increased tumor cell killing with larger RT fractions and preclinical evidence for synergism between RT and erlotinib.

Our hypothesis is that the addition of erlotinib to RT will result in radiosensitization, therefore increasing the likelihood of local tumor control over RT alone. Maintenance erlotinib upon RT completion will result in further tumor growth inhibition, both systemically and locally, lengthening disease-free survival and overall survival.

All eligible patients will be enrolled, without regard for the EGFR status. The implications of prospectively screening patients for EGFR mutations or gene copy number and how the patients should be selected for subsequent treatment remain to be defined (Janne P et al, 2005; Shepherd f et al, 2005). Therefore, patients will not be excluded from trial participation based on the EGFR testing. The EGFR status will be assessed by the FISH assay in biopsy or resection tissue samples and the test will be performed by a commercial laboratory.

ELIGIBILITY:
Inclusion Criteria:

Patients must fulfill all of the following criteria to be eligible for study entry:

* Patients aged 18 years or older with histologically or cytologically confirmed unresectable or medically inoperable NSCLC and measurable disease.
* Patients with AJC Stage IV (metastatic) NSCLC who need initial thoracic RT to control symptoms such as hemoptysis, airway obstruction, esophageal compression, superior vena cava syndrome, other symptoms, or to prevent symptomatic tumor progression.
* Patients with synchronous brain metastases will be allowed to enroll and to receive whole-brain radiation therapy while on the protocol.
* Patients with unresectable or medically inoperable locally advanced (AJC Stage II, IIIA or IIIB) NSCLC, who require thoracic RT but do not qualify for other protocols due to the presence of a malignant pleural or pericardial effusion, major weight loss, poor performance status, unwillingness to receive chemotherapy or other factors.
* Patients with medically inoperable Stage I NSCLC or those patients with a resectable Stage I NSCLC who decline surgery.
* Patients treated initially with systemic chemotherapy or biologic therapy who eventually develop progression of intrathoracic disease and require thoracic RT, or who may benefit from consolidative thoracic RT following chemotherapy or biologic therapy.
* Patients must have a minimal FEV1 of 1.2 l. Lower FEV1 may be allowed for small tumors and a V17 <25%.
* Estimated life expectancy of 3 months or more.
* Patients able to provide a written informed consent prior to study entry.
* Patients who agree to have their biopsy or surgical specimen analyzed for the EGFR status.
* Women of childbearing potential must be willing to practice acceptable methods of birth control to prevent pregnancy.

Exclusion Criteria:

Any of the following is a criterion for exclusion from the trial:

* Small cell lung cancer, any stage
* Previous thoracic radiation therapy
* Oxygen-dependent patients
* FEV1 < 1.2 l
* Patients with severe underlying lung disease of any origin, which in the opinion of the investigators may markedly increase the risk of treatment-related pneumonitis
* Known severe hypersensitivity to Erlotinib or any of the excipients of this product
* Concomitant use of phenytoin, carbamazepine, barbiturates, rifampicin, phenobarbital, or St John's Wort preparations
* Treatment with a nonapproved or investigational drug within 30 days before Day 1 of trial treatment
* Incomplete healing from previous oncologic or other major surgery
* Serum creatinine level greater than CTC grade 2
* Pregnancy or breast feeding (women of childbearing potential)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-08-27 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Werner-Wasik, MD, Principal Investigator — Thomas Jefferson University
Locations (2):
- United States (2):
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Thomas Jefferson Univeristy, Philadelphia, Pennsylvania

REFERENCES:
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erlotinib and Radiotherapy
Started | 17
Completed | 17
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Erlotinib and Radiotherapy
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Experience Progression-free Survival.
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Erlotinib and Radiotherapy
Number analyzed (Participants) | 17
Participants | 1

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Erlotinib and Radiotherapy
All-Cause Mortality (participants affected / at risk) | 9/17
Serious Adverse Events (participants affected / at risk) | 15/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib and Radiotherapy (N=17)
Death (General disorders) | 9 (9)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Headache (General disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 1 (1)
Severe pain (back) (Musculoskeletal and connective tissue disorders) | 1 (1)
Mucositis/Stomatitis (Gastrointestinal disorders) | 1 (1)
Dyspnea w/ADL (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Sodium, serum-low (Blood and lymphatic system disorders) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Fatigue (General disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Hyperkalemia (Blood and lymphatic system disorders) | 1 (1)
Muscle weakness, generalized (Musculoskeletal and connective tissue disorders) | 1 (1)
Elevated Glucose (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib and Radiotherapy (N=17)
Alkaline Phosphatase (Blood and lymphatic system disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anorexia (Psychiatric disorders) | 2 (2)
Bilirubin Increased (Blood and lymphatic system disorders) | 6 (6)
Blepharitis (Eye disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Creatinine increased (Blood and lymphatic system disorders) | 3 (3)
Decreased hearing in left ear (General disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Dizziness (General disorders) | 1 (1)
Dry eye (Eye disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Dysgeusia (General disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Edema (General disorders) | 2 (2)
Esophagitis (Gastrointestinal disorders) | 3 (3)
dysmorphic nail bed (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 7 (7)
Fever (Immune system disorders) | 1 (1)
Glucose, serum-high (Blood and lymphatic system disorders) | 3 (3)
Headache (General disorders) | 1 (1)
Elevated Heart Rate (Cardiac disorders) | 1 (1)
Elevated Hemoglobin (Blood and lymphatic system disorders) | 4 (4)
Hypocalcemia (Blood and lymphatic system disorders) | 1 (1)
Hypokalemia (Blood and lymphatic system disorders) | 2 (2)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vaginal Infection (Reproductive system and breast disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Magnesium (Blood and lymphatic system disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (General disorders) | 5 (5)
Pain (General disorders) | 3 (3)
Peripheral neuropathy (Nervous system disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 12 (12)
Tremor (Nervous system disorders) | 2 (2)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vaginal dryness and irritation (Reproductive system and breast disorders) | 1 (1)
White Blood Cells in Urine (Renal and urinary disorders) | 1 (1)
Weight loss (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes